CLINICAL TRIAL: NCT01380860
Title: Primary Prevention of Peristomial Hernias Via Parietal Prostheses: a Randomized, Multicentric Study
Brief Title: Primary Prevention of Peristomial Hernias Via Parietal Prostheses
Acronym: GRECCAR 07
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PHRC-N/2011/MP-01; 2011-A01572-39 (Other: ANSM)
Record Dates: First submitted 2011-06-22; First posted 2011-06-27 (Estimated); Last update posted 2025-12-01 (Actual); Status verified 2020-08

CONDITIONS: Parastomal Hernia
Keywords: mesh; hernia
MeSH Terms: conditions — Hernia | interventions — Colostomy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mesh (Experimental): The patients allocated to this arm of the study will have mesh (Covidien France: mono filament polyester bidimensional knit) implanted in association with their colostomy.
  Interventions: Procedure: Colostomy with mesh implantation
- No mesh (Active Comparator): The patients allocated to this arm of the protocol will not receive mesh implantation with their colostomy.
  Interventions: Procedure: Simple colostomy

INTERVENTIONS:
Procedure: Colostomy with mesh implantation — Colostomy with mesh implantation
  Arms: Mesh
Procedure: Simple colostomy — Colostomy with no mesh implantation.
  Arms: No mesh

SUMMARY:
The purpose of this study is to compare rates of hernia formation between colostomies created with no hernia preventing mesh versus colostomies created with a particular mesh.

DETAILED DESCRIPTION:
Previous studies indicate that implanting mesh for peristomal hernia repair may efficiently prevent hernia relapse. However, mesh provides a good infection site, which is not a desirable characteristic for a material adjacent to a colostomy "port". Our goal is to implement a high-quality, randomized trial to demonstrate whether or not systematic mesh implantation upon primary hernia creation is an effective means of avoiding this common and troublesome complication.

ELIGIBILITY:
Inclusion Criteria:

* The patient has given informed consent
* The patient must be affiliated with a health insurance programme
* The patient must be available for 24 months of follow-up
* The patient requires a colostomy (primo-event, ie first colostomies only)

Exclusion Criteria:

* The patient is currently participating in another interventional study
* The patient is in an exclusion period determined by a previous study
* The patient is under guardianship
* The patient refuses to sign the consent
* It is impossible to communicate information to the patient (does not read French)
* The patient is pregnant
* The patient is breastfeeding
* There is a contra-indication for any treatment used in this study
* The subject has already had a colostomy
* The subject has peritonitis
* The subject needs a colostomy for infectious reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-11; Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Presence/absence of a peristomal hernia | 24 months
  The occurrence of peristomal hernias is determined in both groups every three months up until 24 months. The presence of absence of a hernia is detected by clinical exam, and at 24 months by an additional radiology exam. The primary outcome concerns rates at 24 months, primo-events only.

SECONDARY OUTCOMES:
Presence/absence of peristomal hernia | 12 months
  The presence of absence of a hernia is detected by clinical exam.
Days of hospitalisation | 1 month
  The number of days spent in the hospital after the surgical intervention.
Operating time (minutes) | Day 1
Estimation of blood loss during the operation (ml) | Day 1
Was stomal repair necessary for the patient? yes/no | 24 months
Was relocation of the colostomy required? yes/no | 24 months
Presence/absence of complications | 24 months
  Complications include: retraction, stenosis, prolapse, disunion, necrosis, abcess, infections, occlusion, strangulation, perforation, eczema, dermatitis, erythema, ulceration
Patient difficulty for fitting his/her colostomy with the appropriate sac. | 24 months
  A visual analog scale is used to determine how difficult it is for a patient to fit his/her colostomy with an appropriate device. 0: perfect adhesion; 10: the device does not adjust to the shape of my skin, and I have permanent leakage.
Pain around the colostomy | 24 months
  A visual analog scale is used to assess the patient's perception of pain around the stomy site.
Abdominal pain | 24 months
  A visual analog scale is used to assess the patient's perception of abdominal pain.
Pain medication consumption | 24 months
Number of colostomy leaks per day | 24 months
Number of colostomy sac changes per day | 24 months
Does the patient consider fitting a sac to his/her colostomy to be a difficult task? yes/no | 24 months
Questionnaire Stoma-QOL | 24 months
  Validated assessment of quality of life.
Exposition of the prothesis (mesh): yes/no | 24 months
Questionnaire Stoma-QOL | 12 months
  Validated assessment of quality of life.
Questionnaire Stoma-QOL | 1 month
  Validated assessment of quality of life.
Presence/absence of peri-operative complications | Day 1
Pain around the colostomy | Day 1
  A visual analog scale is used to assess the patient's perception of pain around the stomy site.
Pain around the colostomy | 1 month
  A visual analog scale is used to assess the patient's perception of pain around the stomy site.
Pain around the colostomy | 3 months
  A visual analog scale is used to assess the patient's perception of pain around the stomy site.
Pain around the colostomy | 6 months
  A visual analog scale is used to assess the patient's perception of pain around the stomy site.
Pain around the colostomy | 9 months
  A visual analog scale is used to assess the patient's perception of pain around the stomy site.
Pain around the colostomy | 12 months
  A visual analog scale is used to assess the patient's perception of pain around the stomy site.
Pain around the colostomy | 15 months
  A visual analog scale is used to assess the patient's perception of pain around the stomy site.
Pain around the colostomy | 18 months
  A visual analog scale is used to assess the patient's perception of pain around the stomy site.
Pain around the colostomy | 21 months
  A visual analog scale is used to assess the patient's perception of pain around the stomy site.
Abdominal pain | Day 1
  A visual analog scale is used to assess the patient's perception of abdominal pain.
Abdominal pain | 1 month
  A visual analog scale is used to assess the patient's perception of abdominal pain.
Abdominal pain | 3 months
  A visual analog scale is used to assess the patient's perception of abdominal pain.
Abdominal pain | 6 months
  A visual analog scale is used to assess the patient's perception of abdominal pain.
Abdominal pain | 9 months
  A visual analog scale is used to assess the patient's perception of abdominal pain.
Abdominal pain | 12 months
  A visual analog scale is used to assess the patient's perception of abdominal pain.
Abdominal pain | 15 months
  A visual analog scale is used to assess the patient's perception of abdominal pain.
Abdominal pain | 18 months
  A visual analog scale is used to assess the patient's perception of abdominal pain.
Abdominal pain | 21 months
  A visual analog scale is used to assess the patient's perception of abdominal pain.
Presence/absence of peristomal hernia | 1 month
  The presence of absence of a hernia is detected by clinical exam.
Presence/absence of peristomal hernia | 3 months
  The presence of absence of a hernia is detected by clinical exam.
Presence/absence of peristomal hernia | 6 months
  The presence of absence of a hernia is detected by clinical exam.
Presence/absence of peristomal hernia | 9 months
  The presence of absence of a hernia is detected by clinical exam.
Presence/absence of peristomal hernia | 15 months
  The presence of absence of a hernia is detected by clinical exam.
Presence/absence of peristomal hernia | 18 months
  The presence of absence of a hernia is detected by clinical exam.
Presence/absence of peristomal hernia | 21 months
  The presence of absence of a hernia is detected by clinical exam.
Presence/absence of complications | 1 month
  Complications include: retraction, stenosis, prolapse, disunion, necrosis, abcess, infections, occlusion, strangulation, perforation, eczema, dermatitis, erythema, ulceration
Presence/absence of complications | 3 months
  Complications include: retraction, stenosis, prolapse, disunion, necrosis, abcess, infections, occlusion, strangulation, perforation, eczema, dermatitis, erythema, ulceration
Presence/absence of complications | 6 months
  Complications include: retraction, stenosis, prolapse, disunion, necrosis, abcess, infections, occlusion, strangulation, perforation, eczema, dermatitis, erythema, ulceration
Presence/absence of complications | 9 months
  Complications include: retraction, stenosis, prolapse, disunion, necrosis, abcess, infections, occlusion, strangulation, perforation, eczema, dermatitis, erythema, ulceration
Presence/absence of complications | 12 months
  Complications include: retraction, stenosis, prolapse, disunion, necrosis, abcess, infections, occlusion, strangulation, perforation, eczema, dermatitis, erythema, ulceration
Presence/absence of complications | 15 months
  Complications include: retraction, stenosis, prolapse, disunion, necrosis, abcess, infections, occlusion, strangulation, perforation, eczema, dermatitis, erythema, ulceration
Presence/absence of complications | 18 months
  Complications include: retraction, stenosis, prolapse, disunion, necrosis, abcess, infections, occlusion, strangulation, perforation, eczema, dermatitis, erythema, ulceration
Presence/absence of complications | 21 months
  Complications include: retraction, stenosis, prolapse, disunion, necrosis, abcess, infections, occlusion, strangulation, perforation, eczema, dermatitis, erythema, ulceration
Patient difficulty for fitting his/her colostomy with the appropriate sac. | Day 1
  A visual analog scale is used to determine how difficult it is for a patient to fit his/her colostomy with an appropriate device. 0: perfect adhesion; 10: the device does not adjust to the shape of my skin, and I have permanent leakage.
Patient difficulty for fitting his/her colostomy with the appropriate sac. | 1 month
  A visual analog scale is used to determine how difficult it is for a patient to fit his/her colostomy with an appropriate device. 0: perfect adhesion; 10: the device does not adjust to the shape of my skin, and I have permanent leakage.
Patient difficulty for fitting his/her colostomy with the appropriate sac. | 3 months
  A visual analog scale is used to determine how difficult it is for a patient to fit his/her colostomy with an appropriate device. 0: perfect adhesion; 10: the device does not adjust to the shape of my skin, and I have permanent leakage.
Patient difficulty for fitting his/her colostomy with the appropriate sac. | 6 months
  A visual analog scale is used to determine how difficult it is for a patient to fit his/her colostomy with an appropriate device. 0: perfect adhesion; 10: the device does not adjust to the shape of my skin, and I have permanent leakage.
Patient difficulty for fitting his/her colostomy with the appropriate sac. | 9 months
  A visual analog scale is used to determine how difficult it is for a patient to fit his/her colostomy with an appropriate device. 0: perfect adhesion; 10: the device does not adjust to the shape of my skin, and I have permanent leakage.
Patient difficulty for fitting his/her colostomy with the appropriate sac. | 12 months
  A visual analog scale is used to determine how difficult it is for a patient to fit his/her colostomy with an appropriate device. 0: perfect adhesion; 10: the device does not adjust to the shape of my skin, and I have permanent leakage.
Patient difficulty for fitting his/her colostomy with the appropriate sac. | 15 months
  A visual analog scale is used to determine how difficult it is for a patient to fit his/her colostomy with an appropriate device. 0: perfect adhesion; 10: the device does not adjust to the shape of my skin, and I have permanent leakage.
Patient difficulty for fitting his/her colostomy with the appropriate sac. | 18 months
  A visual analog scale is used to determine how difficult it is for a patient to fit his/her colostomy with an appropriate device. 0: perfect adhesion; 10: the device does not adjust to the shape of my skin, and I have permanent leakage.
Patient difficulty for fitting his/her colostomy with the appropriate sac. | 21 months
  A visual analog scale is used to determine how difficult it is for a patient to fit his/her colostomy with an appropriate device. 0: perfect adhesion; 10: the device does not adjust to the shape of my skin, and I have permanent leakage.
Pain medication consumption | Day 1
Pain medication consumption | 1 month
Pain medication consumption | 3 months
Pain medication consumption | 6 months
Pain medication consumption | 9 months
Pain medication consumption | 12 months
Pain medication consumption | 15 months
Pain medication consumption | 18 months
Pain medication consumption | 21 months
Number of colostomy leaks per day | Day 1
Number of colostomy leaks per day | 1 month
Number of colostomy leaks per day | 3 months
Number of colostomy leaks per day | 6 months
Number of colostomy leaks per day | 9 months
Number of colostomy leaks per day | 12 months
Number of colostomy leaks per day | 18 months
Number of colostomy leaks per day | 15 months
Number of colostomy leaks per day | 21 months
Number of colostomy sac changes per day | Day 1
Number of colostomy sac changes per day | 1 month
Number of colostomy sac changes per day | 3 months
Number of colostomy sac changes per day | 6 months
Number of colostomy sac changes per day | 9 months
Number of colostomy sac changes per day | 12 months
Number of colostomy sac changes per day | 15 months
Number of colostomy sac changes per day | 18 months
Number of colostomy sac changes per day | 21 months
Does the patient consider fitting a sac to his/her colostomy to be a difficult task? yes/no | Day 1
Does the patient consider fitting a sac to his/her colostomy to be a difficult task? yes/no | 1 month
Does the patient consider fitting a sac to his/her colostomy to be a difficult task? yes/no | 3 months
Does the patient consider fitting a sac to his/her colostomy to be a difficult task? yes/no | 6 months
Does the patient consider fitting a sac to his/her colostomy to be a difficult task? yes/no | 9 months
Does the patient consider fitting a sac to his/her colostomy to be a difficult task? yes/no | 12 months
Does the patient consider fitting a sac to his/her colostomy to be a difficult task? yes/no | 15 months
Does the patient consider fitting a sac to his/her colostomy to be a difficult task? yes/no | 18 months
Does the patient consider fitting a sac to his/her colostomy to be a difficult task? yes/no | 21 months
Exposition of the prothesis (mesh): yes/no | 1 month
Exposition of the prothesis (mesh): yes/no | 3 months
Exposition of the prothesis (mesh): yes/no | 6 months
Exposition of the prothesis (mesh): yes/no | 9 months
Exposition of the prothesis (mesh): yes/no | 12 months
Exposition of the prothesis (mesh): yes/no | 15 months
Exposition of the prothesis (mesh): yes/no | 18 months
Exposition of the prothesis (mesh): yes/no | 21 months
Presence/absence of a complication potentially linked to the presence of a mesh? | 1 month
Presence/absence of a complication potentially linked to the presence of a mesh? | 3 months
Presence/absence of a complication potentially linked to the presence of a mesh? | 6 months
Presence/absence of a complication potentially linked to the presence of a mesh? | 9 months
Presence/absence of a complication potentially linked to the presence of a mesh? | 12 months
Presence/absence of a complication potentially linked to the presence of a mesh? | 15 months
Presence/absence of a complication potentially linked to the presence of a mesh? | 18 months
Presence/absence of a complication potentially linked to the presence of a mesh? | 21 months
Presence/absence of a complication potentially linked to the presence of a mesh? | 24 months
Ablation of the mesh: yes/no | 1 month
Ablation of the mesh: yes/no | 3 months
Ablation of the mesh: yes/no | 6 months
Ablation of the mesh: yes/no | 9 months
Ablation of the mesh: yes/no | 12 months
Ablation of the mesh: yes/no | 15 months
Ablation of the mesh: yes/no | 18 months
Ablation of the mesh: yes/no | 21 months
Ablation of the mesh: yes/no | 24 months
Evaluation of colostomy healing by the clinician | Day 1
  The evaluating clinician (blind to the procedure) will evaluate the healing progress of the colostomy using a visual analog scale.
Evaluation of colostomy healing by the clinician | 1 month
  The evaluating clinician (blind to the procedure) will evaluate the healing progress of the colostomy using a visual analog scale.
Evaluation of colostomy healing by the clinician | 3 months
  The evaluating clinician (blind to the procedure) will evaluate the healing progress of the colostomy using a visual analog scale.
Evaluation of colostomy healing by the clinician | 6 months
  The evaluating clinician (blind to the procedure) will evaluate the healing progress of the colostomy using a visual analog scale.
Evaluation of colostomy healing by the clinician | 9 months
  The evaluating clinician (blind to the procedure) will evaluate the healing progress of the colostomy using a visual analog scale.
Evaluation of colostomy healing by the clinician | 12 months
  The evaluating clinician (blind to the procedure) will evaluate the healing progress of the colostomy using a visual analog scale.
Evaluation of colostomy healing by the clinician | 15 months
  The evaluating clinician (blind to the procedure) will evaluate the healing progress of the colostomy using a visual analog scale.
Evaluation of colostomy healing by the clinician | 18 months
  The evaluating clinician (blind to the procedure) will evaluate the healing progress of the colostomy using a visual analog scale.
Evaluation of colostomy healing by the clinician | 21 months
  The evaluating clinician (blind to the procedure) will evaluate the healing progress of the colostomy using a visual analog scale.
Evaluation of colostomy healing by the clinician | 24 months
  The evaluating clinician (blind to the procedure) will evaluate the healing progress of the colostomy using a visual analog scale.
Duration of postoperative fever (hours) | 10 days
Presence/absence of postoperative fever > 37.2°C | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Michel Prudhomme, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (22):
- France (22):
  - CHRU de Besancon, Besançon
  - CHU de Bordeaux, Bordeaux
  - CHRU de Clermont Ferrand, Clermont-Ferrand
  - APHP - Hôpital Beaujon, Clichy
  - Hôpital Albert Michallon, CHU de Grenoble, Grenoble
  - APHP - Centre Hospitalier Universitaire de Bicêtre, Le Kremlin-Bicêtre
  - Centre de Lutte Contre le Cancer - Centre Oscar Lambret, Lille
  - CHRU de Lille - Hôpital Claude Huriez, Lille
  - CHU de Lyon, Lyon
  - Centre Régional de Lutte Contre le Cancer - Institut Paoli-Calmettes, Marseille
  - APHM - Hôpital La Timone Adultes, Marseille
  - Centre Régional de Lutte Contre le Cancer Val d'Aurelle - Paul Lamarque, Montpellier
  - CHU de Nantes, Nantes
  - Centre Hospitalier Universitaire de Nîmes, Nîmes
  - APHP - Hôpital Lariboisière, Paris
  - APHP - Hôpital Saint-Antoine, Paris
  - APHP - Groupe Hospitalier Pitié-Salpetrière, Paris
  - Hôpital Pontchailou, Rennes
  - CHU de Rouen, Rouen
  - Centre Régional de Lutte contre le Cancer Centre Paul Strauss, Strasbourg
  - CHU de Toulouse, Toulouse
  - CH de Vichy - Jacques Larin, Vichy

REFERENCES:
- [Result] Prudhomme M, Rullier E, Lakkis Z, Cotte E, Panis Y, Meunier B, Rouanet P, Tuech JJ, Jafari M, Portier G, Dubois A, Sielezneff I, Parc Y, Faucheron JL, Meurette G, Lelong B, Piessen G, Karoui M, Fabbro-Peray P, Demattei C, Bertrand MM; GRECCAR research group. End Colostomy With or Without Mesh to Prevent a Parastomal Hernia (GRECCAR 7): A Prospective, Randomized, Double Blinded, Multicentre Trial. Ann Surg. 2021 Dec 1;274(6):928-934. doi: 10.1097/SLA.0000000000004371. PMID 33201089
- [Derived] Prudhomme M, Alline M, Chauvat J, Fabbro-Perray P, Ripoche J, Bertrand MM; French Research Group of Rectal Cancer Surgery (GRECCAR). Primary prevention of peristomial hernias via parietal prostheses: A randomized, multicentric study (GRECCAR 7 trial). Dig Liver Dis. 2016 Jul;48(7):812-6. doi: 10.1016/j.dld.2016.03.020. Epub 2016 Apr 5. PMID 27130912